CLINICAL TRIAL: NCT00553982
Title: Patellar Resurfacing in Total Knee Arthroplasty. A Prospective, Randomised and Double Blind Study.
Brief Title: Patellar Resurfacing in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Eirik Aunan, MD, Sykehuset Innlandet HF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aue1; 40-07172b 1.2007.952 (REK); 13-2007 SI (Personvernombudet)
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis; Pain
Keywords: Replacement; Knee; Patella; Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Pain; Patella Fracture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Patellar resurfacing
  Interventions: Procedure: Patellar component
- 2 (Active Comparator): Patellar retention
  Interventions: Procedure: No patellar component

INTERVENTIONS:
Procedure: Patellar component — Resurfacing with onlay technique
  Arms: 1
Procedure: No patellar component — Trimming of osteophytes when appropriate
  Arms: 2

SUMMARY:
Background:

The best treatment of the patella during total knee arthroplasty (TKA) is controversial. The implantation of a patellar component adds to the operation time and the costs of the operation.There is a huge variation as to whether the patella is resurfaced or not during TKA. Meta-analysis of prospective, randomised trials might indicate that patellar resurfacing reduces the risk of reoperation and anterior knee pain, but drawing firm conclusions is not possible and additional, high quality randomised trials are required.

Purpose:

The aim of this study is to determine whether ther is a difference between the two groups in knee pain, functions, patient satisfaction and quality of life after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 85 years old with osteoarthritis scheduled for primary knee arthroplasty.

Exclusion Criteria:

* Patients who are not able to cooperate
* Serious deformity (not suitable for a standard CR prosthesis)
* Patellar thickness less than 18 mm
* Prior operation involving the extensor mechanism
* Rheumatoid arthritis
* Severe medical disability limiting the ability to walk
* Revision surgery
* Knees with predominantly patellofemoral arthrosis

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-10; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | 3 years follow up

SECONDARY OUTCOMES:
Oxford score, Knee Society score, Stair climbing test, Pain (VAS), Patient satisfaction (VAS) | 3 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Aunan, Doctor, Principal Investigator — Sykehuset Innlandet, Lillehammer
Locations (1):
- Sykehuset Innlandet HF, Lillehammer, Lillehammer, Norway